CLINICAL TRIAL: NCT04346069
Title: Role Of Parent-Child Interaction Therapy Towards Management Of Language And Behavioral Problems Among Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Isra University (Other)
Responsible Party: Principal Investigator, Shahnaz, Principal Investigator, Isra University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IsraUP
Record Dates: First submitted 2020-03-14; First posted 2020-04-15 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Disorder of Speech and Language Development

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regular speech therapy (Other): Regular speech therapy will be provided to the controlled group
  Interventions: Other: PCIT (parent child interaction therapy)
- Parent-child interaction therapy (Other): Parent child interaction therapy will be provided to the experimental group
  Interventions: Other: PCIT (parent child interaction therapy)

INTERVENTIONS:
Other: PCIT (parent child interaction therapy) — Parent child interaction therapy is a treatment strategy that nurture parent child relationship and teach effective parenting strategies to decrease child non compliance behavior (BodifordMcNeil; Hembree-Kigin, 2010).Parent-Child Interaction Therapy (PCIT; Eyberg; Robinson, 1982 ; Zisser; Eyberg, 2008 ) is a manualized parent training intervention that has received substantial empirical support in the treatment of disruptive behavior across multiple reviews (e.g., Brestan; Eyberg, 1998 ; Gallagher, 2003 ; Thomas & Zimmer-Gembeck, 2007 ). PCIT established strong relation among parenting, social learning, and attachment theories and proceeds.
  Other Names: Regular speech therapy

SUMMARY:
maltreatment are particularly vulnerable towards child abuse and developing mental and physical health issues.

parent child interaction therapy (PCIT)) is one of those interventions which can address these vulnerabilities by improving parent to child relation and interaction, primarily improving parenting skills and helping parents cope with their parenting stress and child's behavioral problems.

PCIT is empirically validated to decrease parenting stress, couple conflict and enhance parent child interaction, resulting in better coping skills while parenting for a child with disability.

This research is very vital as it measures the efficacy of parent child interaction.

In Pakistan mostly parents are bringing their children to clinic without any support from government therefore it is not possible for everyone to get daily based therapeutic intervention.

The area of Parent-child Interaction Therapy and the acceptance of these treatments are new and emerging in Pakistani Health Care, apart from above; this research will also assist in identifying further areas of research.

DETAILED DESCRIPTION:
The objective of this study is to determine the efficacy of parent-based intervention in Pakistan.

Parent-Child Interaction Therapy PCIT in treating the behavior problem and language problem due to behavioral disturbances in young children more than usual treatments.

1. To assess efficacy of PCIT intervention program.
2. To translate the Eyeberg Child Behavior Inventory (ECBI), Child-Parent Relationship Scale, Child Behavior Checklist (CBCL) , Test of Early Language-3rd edition (TELD-3) and applications in Urdu language.
3. To translate Child-Parent Relationship Scale and applications in Urdu language.
4. To translate Child Behavior Checklist (CBCL) and applications in Urdu language.
5. To translate Test of Early Language-3rd edition (TELD-3) and applications in Urdu language.
6. To translate parenting relation questionnaire (PQR) in Urdu language.
7. To translate parent stress index (PSI) in Urdu.
8. To determine the reliability and validity of the Urdu translated interventional and assessment tools.
9. To determine prior to and at the conclusion of the intervention performance on measures of parenting relation, parenting tress, children compliance.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for children:

* Participants of the study age between 2to 7years however both the genders are included
* Referred cases for language delay, behavioral or attention/hyperactive problems
* ECBI score of greater than 120
* Parental consent to the study

Inclusion Criteria for Parents:

* Biological Parents
* Minimum education: high school
* Willing to participate

Exclusion Criteria:

Exclusion Criteria for children:

* Mental retardation or pervasive developmental disorder in the child.
* Should not be under any other kind of the therapeutical intervention .

Exclusion Criteria for Parents:

* Psychosis or serious drug abuse in parents
* Lack of sufficient proficiency in parents to fill in the questionnaires

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
efficacy of parent chlid interaction therapy (PCIT) | 6 months
  parent child interaction therapy (PCIT)) is one of those interventions which can address these vulnerabilities by improving parent to child relation and interaction, primarily improving parenting skills and helping parents cope with their parenting stress and child's behavioral problems. efficacy will be assessed by the Parenting Stress Index - Short Form
efficacy of parent chlid interaction therapy (PCIT) will be assessed by the Marital Status Inventory | 6 months
efficacy of parent chlid interaction therapy (PCIT) will be assessed by the Child-Parent Relationship Scale . | 6 months
efficacy of parent chlid interaction therapy (PCIT) will be assessed by the Eyeburg inventory. | 6 months